CLINICAL TRIAL: NCT04077424
Title: Single Cell Molecular Analysis of Influenza Vaccine Induced T Cell Responses in Adults 65 Years of Age or Older
Brief Title: Senescent Immunity in Elders and Vaccine Responses (SILVER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Spyros Kalams, Associate Professor Infectious Disease, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: single cell
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Flu Vaccine
Keywords: adult 65 and older
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluad vaccine; Vaccines

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is an open label trial, the study nurse and participant know which of 3 FDA approved influenza vaccines are given (Fluzone-HD, FluAd, or Flublok). However the investigator and outcomes assessor are blinded to the actual vaccine given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fluzone-High Dose (Active Comparator): FDA approved high dose inactivated influenza vaccine (HD-Fluzone)
  Interventions: Biological: Fluzone-High Dose Quadrivalent
- Fluad (Active Comparator): Adjuvanted (MF59) inactivated influenza vaccine (Fluad)
  Interventions: Biological: Fluad
- Recombinant Hemagglutinin vaccine (Flublok) (Active Comparator): Recombinant hemagglutinin vaccine
  Interventions: Biological: Flublock

INTERVENTIONS:
Biological: Fluzone-High Dose Quadrivalent — Seasonal influenza vaccination with FDA approved vaccines for this age group.
  Other Names: High-dose flu vaccine
  Arms: Fluzone-High Dose
Biological: Fluad — Adjuvanted (MF59) inactivated influenza vaccine
  Other Names: standard-dose, inactivated influenza (flu) vaccine
  Arms: Fluad
Biological: Flublock — Recombinant hemagglutinin vaccine
  Other Names: Recombinant Hemagglutinin vaccine
  Arms: Recombinant Hemagglutinin vaccine (Flublok)

SUMMARY:
To study the effects of age on the immune system's response to flu vaccine and to study the connection between the immune system and physical and cognitive changes associated with aging.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and over
* Independent Living (including Assisted Living)

Exclusion Criteria:

* Unable to understand the consent or the study.
* Allergic to any vaccine components, excluding eggs.
* History of Guillain-Barre.
* Residing in a long -term care facility such as a nursing home.

Ages: 65 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kalams, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All relevant findings will be published in peer-reviewed journals and data generated will be presented at national and international meetings. research articles will be deposited in the NIH National Library of Medicine's PubMed Central upon acceptance for publication.
Access Criteria: All relevant findings will be published in peer-reviewed journals and data generated will be presented at national and international meetings. Research articles will be deposited in the NIH National Library of Medicine's PubMed Central upon acceptance for publication. To the extent possible,we will make raw data available in publications (directly or online appendices). If novel techniques are developed and validated, these methods will be shared with the general scientific community in a timely fashion, and also made available via the protocols.io open access platform. As suggested by the NIH , this will be no later than the acceptance for publication of the main findings from the final data set generated within this proposal. If requests for access to data beyond that in our publications are made by members of the scientific community, we will ask that users submit requests for specific analyses, and we will strive to meet all reasonable requests.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluzone-High Dose | Fluad | Recombinant Hemagglutinin Vaccine (Flublok)
Started | 2 | 2 | 6
Completed | 2 | 2 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone-High Dose | Fluad | Recombinant Hemagglutinin Vaccine (Flublok) | Total
Number analyzed (Participants) | 2 | 2 | 6 | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 67.1 (1.6) | 70.5 (2.4) | 72.1 (5.1) | 69.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 1 | 1 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 6 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutinin Antigen Inhibition Assay Titers at Baseline
Description: 2 fold dilution series of serum, and measurement of titer which inhibits hemagglutination.
  Titers were measured for each of 4 antigens in the vaccine (A/Brisbane/2018 (H1N1), A/Kansas/2017 (H3N2), B/Colorado/2017 (Vic), B/Phuket/2013 (Yam))
Time Frame: Baseline Baseline
Population: 1 person in Fluzone HD group received vaccine, but did not return for subsequent visits, so titers were not performed for this participant.
Measure: Median (Inter-Quartile Range); unit: antibody titers
Arm/Group | Fluzone-High Dose | Fluad | Recombinant Hemagglutinin Vaccine (Flublok)
Number analyzed (Participants) | 2 | 2 | 6
antibody titers
  A/Brisbane/2018 (H1N1): number analyzed (Participants) | 1 | 2 | 6
  A/Brisbane/2018 (H1N1) | 20 [20 to 20] | 160 [160 to 160] | 25 [10 to 50]
  A/Kansas/2017 (H3N2): number analyzed (Participants) | 1 | 2 | 6
  A/Kansas/2017 (H3N2) | 40 [40 to 40] | 90 [20 to 160] | 50 [10 to 160]
  B/Colorado/2017 (Vic): number analyzed (Participants) | 1 | 2 | 6
  B/Colorado/2017 (Vic) | 160 [160 to 160] | 240 [160 to 320] | 120 [70 to 200]
  B/Phuket/2013 (Yam): number analyzed (Participants) | 1 | 2 | 6
  B/Phuket/2013 (Yam) | 320 [320 to 320] | 160 [160 to 160] | 100 [35 to 280]

2. Primary Outcome: Hemagglutinin Antigen Inhibition Assay Titers at Day 28
Description: as for outcome 1
Time Frame: Day 28 Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: antibody titers
Arm/Group | Fluzone-High Dose | Fluad | Recombinant Hemagglutinin Vaccine (Flublok)
Number analyzed (Participants) | 2 | 2 | 6
antibody titers
  A/Brisbane/2018 (H1N1): number analyzed (Participants) | 1 | 2 | 6
  A/Brisbane/2018 (H1N1) | 320 [320 to 320] | 120 [70 to 440] | 480 [320 to 640]
  A/Kansas/2017 (H3N2): number analyzed (Participants) | 1 | 2 | 6
  A/Kansas/2017 (H3N2) | 2560 [2560 to 2560] | 160 [160 to 160] | 320 [280 to 1120]
  B/Colorado/2017 (Vic): number analyzed (Participants) | 1 | 2 | 6
  B/Colorado/2017 (Vic) | 640 [640 to 640] | 320 [140 to 560] | 480 [320 to 640]
  B/Phuket/2013 (Yam): number analyzed (Participants) | 1 | 2 | 6
  B/Phuket/2013 (Yam) | 320 [320 to 320] | 160 [160 to 160] | 240 [140 to 640]

ADVERSE EVENTS:
Time Frame: Baseline to day 28
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion.
Arm/Group | Fluzone-High Dose | Fluad | Recombinant Hemagglutinin Vaccine (Flublok)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT04077424/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04077424/ICF_001.pdf